CLINICAL TRIAL: NCT07128056
Title: Effect of Mobile Phone Video Games on Preoperative Anxiety and Postoperative Pain in Children Undergoing Elective Surgery
Brief Title: Effect of Mobile Phone Video Games on Preoperative Anxiety and Postoperative Pain in Children
Acronym: VAPiC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Numeri (Other Government)
Collaborators: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Sponsor-Investigator, Fatima Numeri, Professor of Paediatric surgery, Services Institute of Medical Sciences, Pakistan
Organization: Services Institute of Medical Sciences, Pakistan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PEDS-ANXPAIN-2025-01; IRB/2024/1434/SIMS (Other: Services Institute of Medical Sciences Lahore,Pakistan)
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Preoperative Anxiety; Postoperative Pain; Elective Surgical Procedure
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-group trial in which pediatric patients undergoing elective surgery will be allocated in a 1:1 ratio to either the intervention arm, receiving mobile phone video game play in addition to standard perioperative care, or the control arm, receiving standard perioperative care alone. Both groups will be assessed for preoperative anxiety and postoperative pain using validated pediatric scales at specified time points.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors who score preoperative anxiety (m-YPAS-SF) and postoperative pain (Wong-Baker FACES) will be blinded to participants' group assignment. Clinical staff and participants cannot be blinded due to the nature of the intervention (mobile phone video games). Assessors will be instructed not to ask about the intervention, and data collection will use standardized forms. The statistician performing primary analyses will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile phone video game distraction (Experimental): Participants will play age-appropriate, non-violent mobile phone video games for approximately 20 minutes before induction of anesthesia as a distraction technique, in addition to receiving standard perioperative care
  Interventions: Behavioral: Mobile phone video game distraction; Other: Standard peri operative care
- Standard perioperative care (Active Comparator): Participants will receive standard perioperative care according to institutional protocols, without exposure to the mobile phone video game distraction
  Interventions: Other: Standard peri operative care

INTERVENTIONS:
Behavioral: Mobile phone video game distraction — Children in the intervention group will play age-appropriate, non-violent mobile phone video games for approximately 20 minutes before induction of anesthesia. This is intended as a distraction technique to reduce preoperative anxiety and improve postoperative pain outcomes. Participants will also receive standard perioperative care.
  Arms: Mobile phone video game distraction
Other: Standard peri operative care — Standard preoperative and postoperative care according to institutional protocol, without mobile phone video game distraction.

SUMMARY:
This randomized controlled trial will evaluate the effect of mobile phone video game distraction on preoperative anxiety and postoperative pain in pediatric surgical patients. Children aged 3-12 years undergoing elective surgery under general anesthesia will be randomly assigned to either a video game distraction group or a control group receiving standard perioperative care. The primary outcomes are preoperative anxiety levels and postoperative pain scores. The study aims to determine whether a simple, low-cost behavioral intervention can improve perioperative experiences in children

DETAILED DESCRIPTION:
Preoperative anxiety and postoperative pain are common problems among pediatric patients undergoing surgery. Children often experience high levels of anxiety before a surgical procedure, and this preoperative anxiety can have long-term negative outcomes. Surgical tissue damage leads to moderate to severe postoperative pain, and preoperative anxiety is a significant predictor of postoperative pain. Inadequate pain management can result in delayed recovery, diminished quality of life, increased healthcare costs, and higher healthcare utilization.

Both pharmacological and non-pharmacological methods are used to manage preoperative anxiety and postoperative pain. However, pharmacological medications may have undesirable side effects, and non-pharmacological interventions such as music therapy, clown presence, or parental presence may not be feasible in the operating theatre environment.

Video games (VGs) are increasingly used in healthcare as distraction tools and for behavior modification therapy. Mobile phones are widely available, and playing video games has become a common activity in society. Children can become deeply engaged in playing VGs, which may reduce their awareness of the surgical environment and lower their anxiety levels. Reduced preoperative anxiety may, in turn, lead to decreased postoperative pain.

There is a lack of local research on the use of mobile phone video games in pediatric perioperative care. This study aims to evaluate the effect of mobile phone video games in reducing preoperative anxiety and postoperative pain, and to determine whether this intervention can be recommended for pediatric surgeries.

A randomized controlled trial will be conducted in the Department of Pediatric Surgery, Services Hospital Lahore, over 12 months. Children aged 3-12 years undergoing low-risk elective surgery will be enrolled. Informed consent will be obtained from parents or guardians. Participants will be randomized via the lottery method into:

* Experimental group: Mobile phone video game distraction (n=75)
* Control group: Standard perioperative care (n=75)

Anxiety will be measured at two points:

* T1: In the preoperative waiting room
* T2: After playing video games for 20 minutes, before induction of anesthesia in the operating room

The Modified Yale Preoperative Anxiety Scale - Short Form (m-YPAS-SF) will be used, where scores range from 22.92 to 100, with lower scores indicating lower anxiety. Postoperative pain will be assessed in the ward using the Revised Faces Pain Scale (r-FACES).

Data will be analyzed using SPSS v25. Numerical variables will be summarized as mean ± standard deviation, and categorical variables as frequencies and percentages. Independent sample t-tests will be used for numerical variables, and Chi-square tests for categorical variables. Data will be stratified for age, gender, and weight to control for effect modifiers. A p-value ≤ 0.05 will be considered statistically significant.

Preoperative anxiety management is a relatively neglected area in Pakistan, and international recommendations are not always applicable in resource-limited settings. The findings from this single-center clinical trial will provide evidence for local clinical practice and may serve as a framework for developing regional protocols to prevent adverse postoperative outcomes.

Limitations: Single-center design and the need for additional staff and time to conduct the study

ELIGIBILITY:
Inclusion Criteria:

* Age 3-12y
* Children undergoing elective surgery
* Has access to a Mobile phone
* Is able to speak in urdu
* Children with no contraindications for the use of video games

Exclusion Criteria:

* Children with previous surgical experience
* Children with cognitive and learning disabilities
* Children with a chronic illness/pain that required special medical care
* Not familiar with video games

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Preoperative Anxiety Level | Measured twice - (T1) in the preoperative waiting area before intervention, and (T2) after 20 minutes of mobile phone video game distraction, immediately before induction of anesthesia.
  Anxiety will be measured at two time points (T1 and T2). At T1, baseline anxiety will be assessed in the preoperative waiting room. Children randomized to the intervention group will then play mobile phone video games for 20 minutes, while the control group will not. At T2, anxiety will be reassessed immediately before induction of anesthesia in the operating room. Anxiety will be measured using the modified Yale Preoperative Anxiety Scale - Short Form (m-YPAS-SF), where scores range from 22.92 to 100, with lower scores indicating lower anxiety.
Postoperative Pain Intensity | It will be measured at 1 and 12 hours after surgery in the ward.
  Post operative pain management will be standardized and it will be measured at 1 and 12 hours after surgery using revised faces pain scale (FPS-r) in the ward.It consists of six faces showing progressively increasing levels of distress with each face assigned a numerical value 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Dr Fatima Naumeri, FCPS,MCPS-HPE,MCPS,CME, Study Director — Services Institute of Medical Sciences, Pakistan
Locations (1):
- Department of Pediatric Surgery ,Services Institute of Medical Sciences/Services Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bezgin S, Kuyulu S, Atıcı A. Investigation of the effect of video-based game application on acute pain in children under surgery. Journal of Health Sciences and Medicine. 2025;8(1):115-118. doi:10.32322/jhsm.123456
- [Background] Teruel J, Stafford G, Brown J, Jones B, Hopkins M, Johnson A, Edenfield J, Guo A, Schammel C, Renfro S, Nisonson A. Reduction of perioperative anxiety using a hand-held video game device: A randomized study. Perioperative Care and Operating Room Management. 2021 Dec;24:100203. doi:10.1016/j.pcorm.2021.100203.
- [Background] Rostami E, Khanjari S, Haghani H, Amirian H. Effect of video games on preoperative anxiety in 3- to-6-year-old of a sample of Iranian children undergoing elective surgery. J Educ Health Promot. 2022 Apr 28;11:135. doi: 10.4103/jehp.jehp_455_21. eCollection 2022. PMID 35677284
- [Background] Mustafa MS, Shafique MA, Zaidi SDEZ, Qamber A, Rangwala BS, Ahmed A, Zaidi SMF, Rangwala HS, Uddin MMN, Ali M, Siddiq MA, Haseeb A. Preoperative anxiety management in pediatric patients: a systemic review and meta-analysis of randomized controlled trials on the efficacy of distraction techniques. Front Pediatr. 2024 Feb 19;12:1353508. doi: 10.3389/fped.2024.1353508. eCollection 2024. PMID 38440185
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] Ali MA, Khan MH, Salim B. Comparing Pharmacological and Nonpharmacological Interventions for Alleviating Preoperative Anxiety in Pediatric Surgical Patients: A Randomized Controlled Trial in Pakistan. Cureus. 2025 Apr 18;17(4):e82502. doi: 10.7759/cureus.82502. eCollection 2025 Apr. PMID 40385813